CLINICAL TRIAL: NCT06028139
Title: Continuous Assessment of Risk and Efficacy (CARE) Using Health Coaching, Continuous Glucose Monitoring and AI Mobile App in Diabetes
Brief Title: Health Coaching, Continuous Glucose Monitoring and AI Mobile App in Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Sengkang General Hospital (Other); National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202208-00017
Record Dates: First submitted 2023-08-28; First posted 2023-09-08 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Continuous glucose monitoring and health coaching; Behavioral: EMPOWER mobile app
- Control (Other)
  Interventions: Behavioral: EMPOWER mobile app

INTERVENTIONS:
Behavioral: Continuous glucose monitoring and health coaching — Each CGM device will work for 14 days. The participants will use the CGM devices for the first two-week period in the first three months of the trial, and the first two-week period of the second three months of the trial.
  Participants will interact with health coach throughout the study duration.
  Arms: Intervention
Behavioral: EMPOWER mobile app — Nudges will be delivered through the EMPOWER mobile app. Participants will log lifestyle information such as diet and physical activity, and clinical information such as medication and HbA1c levels through the EMPOWER mobile app.

SUMMARY:
Lifestyle change is key to diabetes management but there are limited resources and time to support patients in improving lifestyle behaviour in the current healthcare system. Currently, health coaching for behavioural chance guided by continuous glucose data, wearable and lifestyle data is not available in primary and tertiary care management of diabetes. This parallel-group randomised controlled trial (RCT) aims to investigate the effectiveness of a novel multi-component model of care comprising interventions including the mobile app EMPOWER and smartwatch, health coaching, and continuous glucose monitoring (CGM).

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 years and above
* Have diagnosis of type 2 diabetes mellitus
* Provided informed consent
* Have near-field communication (NFC) compatible phones
* Able to engage in light physical activity (e.g., walking)

Exclusion Criteria:

* Significant cognitive impairment
* Other conditions that may preclude participants from wearing CGM devices

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 6 months
  HbA1c over 6 months

SECONDARY OUTCOMES:
Physical activity as measured by number of steps | 6 months
  Physical activity over 6 months
Physical activity as measured by moderate to vigorous active minutes | 6 months
  Physical activity over 6 months
Physical activity as measured by GPAQ | 6 months
  Physical activity over 6 months
Diet as measured by DASH | 6 months
  Diet quality over 6 months
Sugar sweetened beverages intake | 6 months
  Sugar sweetened beverages intake over 6 months
Patient activation score as measured by patient activation measure | 6 months
  Difference in patient activation score between intervention and control over 6 months
Medication adherence as measured by DOSE-Nonadherence scale | 6 months
  Difference in medication adherence between intervention and control over 6 months
Quality of life as measured by EQ-5D-5L | 6 months
  Difference in quality of life between intervention and control over 6 months
Healthcare cost as measured by cost of consultations, lab tests, medications, admission | 6 months
  Healthcare cost over 6 months
Healthcare cost as measured by WPAI | 6 months
  Healthcare cost over 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- Singapore (3):
  - Singapore General Hospital, Singapore
  - National Heart Centre Singapore, Singapore
  - Sengkang General Hospital, Singapore